CLINICAL TRIAL: NCT04149093
Title: The Association Between Calretinin and the Function of Ganglion Cells in Long Segment and Total Hirschsprung Disease
Brief Title: The Association Between Calretinin and the Function of Ganglion Cells in Hirschsprung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Nelson Piche, Principal Investigator, St. Justine's Hospital
Other Study IDs: 2020-2597
Record Dates: First submitted 2019-10-23; First posted 2019-11-04 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hirschsprung Disease; Ganglion; Hirschsprung Disease, Long-Segment; Hypoganglionosis
MeSH Terms: conditions — Hirschsprung Disease; Ganglion Cysts | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Calretinin staining — A paraffin-embedded hematoxylinphloxin-safran sections will be performed on tissue specimens of proximal resection margins to evaluate the presence or absence of ganglion cells.
  Immunohistochemistry (IHC) will then be done on paraffin-embedded sections for calretinin staining.
  Other Names: Immunohistochemistry

SUMMARY:
This study aims to compare the outcomes of patients with long segment Hirschsprung disease or total colonic aganglionosis who had negative calretinin staining and positive ganglion cells on the proximal resection margins to those who had both positive findings.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histopathological diagnosis of Hirschsprung disease from January 1, 1990 to August 31, 2019
* Long-segment Hirschsprung disease (type A and B)
* Total colonic aganglionosis (TCA)
* Surgery at CHUSJ
* Tissue blocks of proximal resection margin available for pathological analysis
* Minimum 1 month of postoperative follow-up

Exclusion Criteria:

* Short-segment Hirschsprung disease (conventional form, rectosigmoid junction)
* Total colonic with small bowel aganglionosis (TCSA)
* Surgery done at another institution
* Early deaths
* Lost to follow-up
* No documented post-operative outcome

Ages: 0 Years to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with Hirschsprung disease and a transition zone more proximal to the distal sigmoid
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Long-term outcomes (Quality of life questionnaire) | 1 year
  To determine if calretinin has a role in the function of ganglion cells in long segment Hirschsprung disease and total colonic aganglionosis.
  HAQL (Hirschsprung's disease and Anorectal malformations Quality of Life) questionnaire. For each item the response is scored from 0 to 3 and then, linearly transformed to a 0 (minimum value) to 100 (maximum value) scale. Higher score suggests a better quality of life.

SECONDARY OUTCOMES:
Surgical complications | 1 year
  * Number of reoperations
  * Number of rebiopsies
  * Number of readmissions
  * Number of bowel obstructions
  * Number of bowel perforation
  * Number of anastomotic leaks
  * Number of anastomotic strictures
  * Number of fistula
  * Number of anal stenosis
  * Number of Hirschsprung-associated enterocolitis
Functional outcomes | 1 year
  * Presence of constipation (yes/no)
  * Presence of diarrhea (yes/no)
  * Presence of incontinence and soiling (yes/no)
  * Presence of abdominal distension (yes/no)
  * Presence of dependance on enemas/medications (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada